CLINICAL TRIAL: NCT03168958
Title: Methadone and Quality of Postoperative Recovery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director Clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH16-374
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Quality of Recovery Scores
MeSH Terms: interventions — Methadone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receieve either methadone or saline-control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drugs will be prepared by the operating room pharmacy. All patients and care providers will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methadone Group (Active Comparator): Patients in this group will receive 0.4 mg/kg of methadone at induction of anesthesia
  Interventions: Drug: Methadone
- Saline-Control Group (Sham Comparator): Patients in this group will receive an equal volume of saline as the active comparator group at induction of anesthesia
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Methadone — Methadone will be provided at induction of anesthesia
  Arms: Methadone Group
Drug: Saline — Saline will be administered at induction of anesthesia
  Arms: Saline-Control Group

SUMMARY:
Patients undergoing cardiac surgery often experience moderate to severe pain in the early postoperative period. A number of methods have been used to help control pain after surgery; however, each of these techniques adds additional costs and risks. A simple and effective way to decrease this pain is to administer a long-acting opioid in the operating room. Methadone is a opioid that can produce analgesia (pain relief) that lasts up to 48 hours when given in large doses (0.3 to 0.4 mg/kg). Previous studies have demonstrated that both pain and requirements for analgesic medications are significantly reduced for up to three days after surgery if methadone is given at induction (the start) of anesthesia. In the study that was performed at Evanston Hospital, cardiac surgical patients who were given methadone also appeared to "feel better" after surgery compared to those given a standard or typical intraoperative opioid. The aim of this randomized clinical trial is to determine whether overall quality of postoperative recovery can be enhanced if methadone is given in the operating room. Quality of recovery will be determined by using a validated scoring system, the QoR 40, which will be given to patients to complete on the first three days after surgery.

DETAILED DESCRIPTION:
Postoperative pain for the adult cardiac surgery patient is complex. Pain can be caused by incisions, intraoperative tissue retraction and dissection, multiple intravascular cannulations, chest tubes left after surgery, and multiple invasive procedures that patients undergo in the operating room and intensive care unit (ICU). Postoperative pain has been described as one of the primary sources of concern for cardiac surgery patients. In this patient population, several studies have demonstrated that pain intensity was moderately severe (approximately 5 on an intensity scale of 10) during the first 2 postoperative days (POD) and did not begin to decline until POD 3. The primary method of pain management used in cardiac surgical patients during early recovery in the intensive care unit (ICU) is the administration of intravenous morphine. Morphine is typically administered per patient request or during nursing assessments for pain. Studies have demonstrated that relatively small doses of morphine (or oral analgesics on the ward) are used following cardiac surgery. The relatively high intensity of postoperative pain and the low doses of analgesics administered suggest that postoperative pain in cardiac surgical patients is an under-recognized and under-treated problem in the early recovery period. Therefore, methods to more successfully manage pain are needed, especially during the first postoperative days.

Opioids remain the primary therapeutic agents for treatment of pain after cardiac surgery. Intermittent (every 3-4 hour) intravenous administration remains the most common mode of delivery. This technique results in significant fluctuations in serum levels of opioids and consequently variability in levels of pain control. An alternative strategy is the use of an opioid with a long half-life which will provide stable blood concentrations after a single intravenous dose. Such an opioid could provide prolonged and constant analgesia. Methadone is an opioid which fulfills these criteria. A primary advantage of methadone is its long half-life, which ranges from 25-52 hours. This unique property of methadone means that single daily doses can be used. Although it is best known as a drug used to treat narcotic addiction, methadone has also been used as an analgesic agent. A number of recent investigations have demonstrated that methadone is effective in treating a number of chronic pain conditions. Methadone has also been studied as an agent to provide prolonged postoperative analgesia. When methadone was administered intravenously to surgical patients, a half-life of 35 hours was observed, resulting in a median duration of analgesia lasting 26 hours. In patients undergoing abdominal, orthopedic, or gynecologic surgery, the use of a single dose of methadone (20 mg or 0.25-0.3 mg/kg) at induction of anesthesia resulted in improved analgesia for the first 24 hours after surgery, when compared to other intraoperative opioids. In these investigations, patients in the methadone groups required significantly less postoperative pain medication and reported lower pain scores during the first postoperative day. Up to 39% of patients required no additional pain medications, despite undergoing major surgery associated with moderate-to severe-levels of postoperative pain. No adverse events directly attributable to methadone were reported in these clinical trials.

Patients undergoing cardiac surgery typically receive a moderate dose of a short-acting opioid (most-commonly fentanyl) at the time of induction of anesthesia. Many clinicians believe that the analgesic effects of fentanyl will persist into the postoperative period. However, when standard doses (500-1000 mcg) of this opioid are given at induction of anesthesia in cardiac patients, a relatively short plasma half-life is observed (3.3 hours). An intraoperative opioid with more desirable pharmacokinetic (long half-life and low clearance) and pharmacodynamic properties may provide for improved postoperative analgesia in a cardiac surgical patient population. In addition to providing for prolonged pain relief, methadone has other unique properties that may be advantageous in cardiac surgical patients. Recent evidence has demonstrated that methadone has the ability to block N-methyl-D-aspartate (NMDA) receptors. NMDA receptors have been implicated in the development of postoperative hyperalgesia (amplification of pain stimuli), and techniques that block NMDA receptors reduce pain. In addition, recent evidence has demonstrated that blockade of NMDA receptors may reduce depression and improve mood. Furthermore, methadone inhibits the reuptake of serotonin and norepinephrine; elevation of these monoamines may play a role in antinociception and mood elevation. Finally, the use of methadone has been reported to be associated with a reduced incidence of nausea and vomiting, when compared to other standard intraoperative opioids. These findings suggest that in addition to providing prolonged and consistent pain relief, methadone may improve several other components of postoperative recovery. Previous studies of opioid use in patients undergoing cardiac surgery have focused on physiologic variables and major adverse events as primary endpoints. As the safety of anesthesia and surgery has improved, assessment of quality of postoperative recovery has become an increasingly important outcome measure in clinical research. Therefore, a comprehensive assessment of postoperative recovery should include factors important to both clinicians (hemodynamic stability, intensive care unit (ICU) length of stay (LOS)) and patients (physical comfort, mood). In particular, an important component of recovery from anesthesia and surgery is patient perception of quality of health in the early postoperative period. Several tools have been recently developed to assess this outcome variable. The QoR-40 is a 40-item scoring system specifically designed to measure health status following anesthesia. The QoR-40 measures five dimensions of recovery: physical comfort (12 questions); emotional state (9 questions); physical independence (5 questions); psychological support (7 questions); and pain (7 questions). Each question is rated by the patient on a five-point Likert scale, with possible scores ranging from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery). A systematic review of instruments used to measure patient-based recovery outcomes determined that the QoR-40 was the only assessment tool that fulfilled the criteria of appropriateness, reliability, validity, responsiveness, precision, interpretability, acceptability, and feasibility. The QoR-40 has been used to assess the impact of anesthetic interventions on recovery after cardiac surgery; furthermore, low postoperative QoR-40 scores have been associated with complications and increased hospital LOS in this patient population.

The primary aim of this randomized, double-blind study is to examine the effect of a single intraoperative dose of methadone on quality of recovery in the early postoperative period. Quality of recovery will be assessed using the QoR 40 scoring system over the first 3 postoperative days. Secondary outcome measures to be assessed will include postoperative pain scores and analgesic requirements, as well as other standard recovery variables (length of postoperative intubation, ICU and hospital length of stay, incidence of nausea or vomiting, level of sedation). Based upon the pharmacokinetic and pharmacodynamics properties of methadone, we hypothesize that patients randomized to receive this long-acting opioid will have improved QoR 40 scores, particularly in the dimensions of physical comfort, emotional state, and pain.

Study Design Patients: One-hundred patients will be enrolled in this clinical trial. All patients presenting for elective cardiac surgery with cardiopulmonary bypass will be eligible for enrollment.

Anesthetic management: Patients will be randomized to receive either methadone or saline-control on the basis of a computer generated random number table. Patients in the methadone group will receive a standard intraoperative dose of methadone that will allow for early tracheal extubation (within 4-8 hours of the conclusion of the surgical procedure). Patients randomized to the methadone group will be given 0.4 mg/kg of methadone at induction of anesthesia (maximal dose 30 mg). Patients assigned to the saline-control group will be administered saline at anesthetic induction. Study drugs will be prepared by the pharmacy. The syringes will be administered over five minutes at induction of anesthesia. The administration of all other anesthetic agents will be standardized and reflect the usual practices of cardiac anesthesiologists at NorthShore. All anesthesia care team members, nurses, surgeons, and researchers will be blinded to group assignment throughout the hospital admission.

Data Collection The primary endpoint of the study is the QoR 40 score. The QoR-40 consists of 40 questions designed to assess quality of recovery following anesthesia and surgery. The QoR 40 will be presented to the patient to complete four times in the perioperative period; immediately before surgery, and the morning (9AM to 11 AM) of postoperative days 1, 2, and 3. The questionnaire will be completed by the patient. If the patient is unable to circle the correct responses on the form, a researcher will verbally present the questions to the patient and then record the responses.

Additional data will be collected by a research assistant at the time the QoR 40 is completed by the patient. Pain on 11-point verbal analogue scale (0=no pain, 10=worst pain imaginable) will be assessed at rest and with coughing. Level of sedation will be determined by observers using a 4-point sedation scale (0=fully awake, 1=mildly sedated (seldom drowsy and easy to awake), 2=moderately sedated (often drowsy and easy to awake), 3=severely sedated (somnolent, difficult to awake). Any episodes of nausea and vomiting will be recorded. Patient satisfaction with overall pain management will be determined using a 100-point verbal rating scale (1=highly dissatisfied (worst), 100=highly satisfied (best)). The amount of pain medication used in each study interval (listed above) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective cardiac surgery with CPB will be eligible for enrollment

Exclusion Criteria:

* Preoperative renal failure requiring dialysis or severe renal dysfunction (serum creatinine > 2.0 mg/dL)
* Significant hepatic dysfunction (liver function tests > 2 times upper normal limit)
* Pulmonary disease necessitating home oxygen therapy
* Preoperative requirement for inotropic agents or intraaortic balloon pump to maintain hemodynamic stability
* Allergy to methadone or fentanyl
* Significant preoperative pain requiring treatment with opioids or recent history of opioid abuse
* Inability to speak or read the English language or neurologic conditions that may impair the ability to complete the QoR 40 questionnaire.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-12-25 (Actual); Primary Completion 2021-05-25 (Estimated); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery scores (QoR 40) on postoperative day 1 | 24 hours
  The QoR 40 scoring system will be used to assess postoperative quality of recovery

SECONDARY OUTCOMES:
Quality of recovery scores (QoR 40) on postoperative day 2 | 48 hours
  The QoR 40 scoring system will be used to assess postoperative quality of recovery
Quality of recovery scores (QoR 40) on postoperative day 3 | 72 hours
  The QoR 40 scoring system will be used to assess postoperative quality of recovery
Pain scores on on postoperative day 1 | 24 hours
  Assessment of pain on 11-point verbal analogue scale (0=no pain, 10=worst pain imaginable)
Pain scores on on postoperative day 1 | 48 hours
  Assessment of pain on 11-point verbal analogue scale (0=no pain, 10=worst pain imaginable)
Analgesic requirements on postoperative day 1 | 24 hours
  The amount of postoperative pain medications will be quantified
Analgesic requirements on postoperative day 2 | 48 hours
  The amount of postoperative pain medications will be quantified
Patient satisfaction scores on postoperative day 1 | 24 hours
  Patient satisfaction with overall pain management will be determined using a 100-point verbal rating scale (1=highly dissatisfied (worst), 100=highly satisfied (best)
Patient satisfaction scores on postoperative day 2 | 48 hours
  Patient satisfaction with overall pain management will be determined using a 100-point verbal rating scale (1=highly dissatisfied (worst), 100=highly satisfied (best)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This data will not be shared with other researchers until publication